CLINICAL TRIAL: NCT03613662
Title: An Open-label, Single-arm Study to Characterize the Pharmacodynamics and Safety of Repeat Dose SP-102 Administered by Epidural Injection in Subjects With Lumbosacral Radiculopathy
Brief Title: A Research Study to Characterize the Pharmacodynamics and Safety of Repeat Dose SP-102
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Semnur Pharmaceuticals, Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other); Scilex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Scilex Pharmaceuticals, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-102-03
Record Dates: First submitted 2018-07-09; First posted 2018-08-03 (Actual); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Lumbosacral Radicular Pain
Keywords: lumbosacral radicular pain; sciatica; leg pain
MeSH Terms: conditions — Sciatica

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SP-102 (Experimental): SP-102
  Interventions: Drug: SP-102

INTERVENTIONS:
Drug: SP-102 — Injection

SUMMARY:
This is an open-label, single-arm, repeat dose study to characterize the pharmacodynamics and safety/tolerability of SP-102 administered by epidural injection.

ELIGIBILITY:
Main Inclusion Criteria:

* Able and willing to read, write, and understand the English language and provide English language written informed consent prior to beginning any study procedures.
* Age 18 to 70 years (inclusive) at the Screening Visit.
* A diagnosis of lumbosacral radicular pain (sciatica).
* Agrees to follow study-specific medication requirements.
* If sexually active and a female of child-bearing potential or a male capable of bearing a child, agrees to use an effective method of birth control during the study.
* Has reviewed all study specific materials and has, in the opinion of the Investigator, the abilities to understand and appropriately complete all study procedures.

Main Exclusion Criteria:

* Has radiologic evidence of a condition that would compromise study outcomes.
* Has ever had lumbosacral back surgery or plans to undergo spine surgical intervention while in the study.
* Has been diagnosed with insulin dependent diabetes mellitus.
* Presence of any other disorder, condition or circumstance (including secondary gain) that, in the opinion of the Investigator, has the potential to prevent study completion and/or to have a confounding effect on outcome assessments.
* Use of any investigational drug and/or device within 30 days, or is scheduled to receive an investigational drug other than blinded study drug during this study.
* Has a body mass index ≥40 kg/m2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Lissin, MD, Study Director — Scilex Pharmaceuticals, Inc.
Locations (1):
- Semnur Research Site 1, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Radnovich R, Heinz J, Ambrose C, Stannard E, Lissin D. Repeat Epidural Injections of SP-102 (Dexamethasone Sodium Phosphate Injectable Gel) in Subjects with Lumbosacral Radiculopathy. J Pain Res. 2021 May 5;14:1231-1239. doi: 10.2147/JPR.S303282. eCollection 2021. PMID 33981160

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SP-102
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SP-102
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (14.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] | 166.51 (12.294)
Weight [Mean (Standard Deviation); unit: kg] | 84.03 (16.412)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.51 (6.127)

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Cortisol Concentrations From Baseline
Description: Dexamethasone-induced hypothalamic-pituitary-adrenal (HPA) suppression is evaluated by monitoring SP-102 induced changes in plasma cortisol levels from Baseline.
  The T1 (index) and T2 (repeat) injections of SP-102 are separated by 4-8 weeks
Time Frame: 12 Weeks
Population: 19 subjects were enrolled and received an index (T1) injection of SP-102. 15 subjects received a (T2) injection of SP-102. Data was not recorded for all subjects at each time point.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | SP-102
Number analyzed (Participants) | 19
nmol/L
  T1: Day 1 (predose) | 36.62 (31.81)
  T1: Day 2: number analyzed (Participants) | 18
  T1: Day 2 | 0.64 (0.27)
  T1: Day 3 | 6.26 (9.00)
  T1: Day 4 | 29.77 (2.60)
  T1: Day 5: number analyzed (Participants) | 18
  T1: Day 5 | 39.91 (40.53)
  T1: Day 8 | 39.71 (28.97)
  T1: Day 15: number analyzed (Participants) | 18
  T1: Day 15 | 44.28 (33.55)
  T1: Day 28 | 25.08 (21.34)
  T2: Day 1 (predose): number analyzed (Participants) | 15
  T2: Day 1 (predose) | 38.81 (41.10)
  T2: Day 2: number analyzed (Participants) | 15
  T2: Day 2 | 0.64 (0.23)
  T2: Day 3: number analyzed (Participants) | 15
  T2: Day 3 | 3.68 (3.85)
  T2: Day 4: number analyzed (Participants) | 15
  T2: Day 4 | 50.71 (56.21)
  T2: Day 5: number analyzed (Participants) | 15
  T2: Day 5 | 38.35 (35.00)
  T2: Day 8: number analyzed (Participants) | 15
  T2: Day 8 | 41.73 (38.95)
  T2: Day 15: number analyzed (Participants) | 14
  T2: Day 15 | 73.31 (97.64)
  T2: Day 28: number analyzed (Participants) | 15
  T2: Day 28 | 28.18 (20.34)

2. Primary Outcome: Change in Blood Glucose Levels From Baseline
Description: Dexamethasone-induced hypothalamic-pituitary-adrenal (HPA) suppression is evaluated by monitoring SP-102 induced changes in blood glucose levels from Baseline.
  The T1 (index) and T2 (repeat) injections of SP-102 are separated by 4-8 weeks
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | SP-102
Number analyzed (Participants) | 19
nmol/L
  T1: Day 1 (predose) | 4.993 (0.5216)
  T1: Day 2 | 6.155 (0.9009)
  T1: Day 3 | 4.528 (0.4451)
  T1: Day 4 | 4.676 (0.5509)
  T1: Day 5: number analyzed (Participants) | 18
  T1: Day 5 | 4.958 (0.4362)
  T1: Day 8 | 5.059 (0.6597)
  T1: Day 15: number analyzed (Participants) | 18
  T1: Day 15 | 5.254 (0.8143)
  T1: Day 28 | 4.963 (0.7116)
  T2: Day 1 (predose): number analyzed (Participants) | 15
  T2: Day 1 (predose) | 4.867 (0.5655)
  T2: Day 2: number analyzed (Participants) | 15
  T2: Day 2 | 5.865 (0.8673)
  T2: Day 3: number analyzed (Participants) | 15
  T2: Day 3 | 4.581 (0.4986)
  T2: Day 4: number analyzed (Participants) | 15
  T2: Day 4 | 4.850 (0.8078)
  T2: Day 5: number analyzed (Participants) | 15
  T2: Day 5 | 4.959 (0.5791)
  T2: Day 8: number analyzed (Participants) | 15
  T2: Day 8 | 4.821 (0.4463)
  T2: Day 15: number analyzed (Participants) | 14
  T2: Day 15 | 5.237 (0.8394)
  T2: Day 28: number analyzed (Participants) | 15
  T2: Day 28 | 4.945 (0.5959)

3. Primary Outcome: Change in White Blood Cell (WBC) Levels From Baseline
Description: Dexamethasone-induced hypothalamic-pituitary-adrenal (HPA) suppression is evaluated by monitoring SP-102 induced changes in WBC levels from Baseline.
  The T1 (index) and T2 (repeat) injections of SP-102 are separated by 4-8 weeks
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cell count × 10^9/L
Arm/Group | SP-102
Number analyzed (Participants) | 19
cell count × 10^9/L
  T1: Day 1 (predose) | 6.65 (2.051)
  T1: Day 2 | 13.43 (3.726)
  T1: Day 3 | 9.33 (2.336)
  T1: Day 4 | 7.38 (1.863)
  T1: Day 5: number analyzed (Participants) | 18
  T1: Day 5 | 6.81 (1.771)
  T1: Day 8 | 6.91 (2.212)
  T1: Day 15: number analyzed (Participants) | 18
  T1: Day 15 | 7.26 (1.873)
  T1: Day 28 | 6.15 (1.339)
  T2: Day 1 (predose): number analyzed (Participants) | 15
  T2: Day 1 (predose) | 6.77 (1.865)
  T2: Day 2: number analyzed (Participants) | 15
  T2: Day 2 | 13.43 (4.517)
  T2: Day 3: number analyzed (Participants) | 15
  T2: Day 3 | 9.21 (3.199)
  T2: Day 4: number analyzed (Participants) | 15
  T2: Day 4 | 7.88 (2.302)
  T2: Day 5: number analyzed (Participants) | 15
  T2: Day 5 | 7.28 (2.087)
  T2: Day 8: number analyzed (Participants) | 14
  T2: Day 8 | 7.31 (2.803)
  T2: Day 15: number analyzed (Participants) | 14
  T2: Day 15 | 8.05 (3.592)
  T2: Day 28: number analyzed (Participants) | 15
  T2: Day 28 | 6.07 (1.541)

4. Secondary Outcome: Change in Numeric Pain Rating Scale (NPRS) Scores for Leg Pain From Baseline
Description: The NPRS is an 11-point scale (0- to 10-point scale where 0 is no pain and 10 is worst pain imaginable) that allows subjects to rate the severity of their pain intensity at various points in time (Turk et al., 2003). Subjects used the NPRS to record their current pain, average pain over 24 hours, and worst pain over 24 hours for both affected leg(s) and back pain. NPRS average leg pain scores over 24 hours are presented.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SP-102
Number analyzed (Participants) | 19
score on a scale
  T1: Baseline (pre-dose) | 5.4 (1.30)
  T1: Day 1 | 5.3 (1.29)
  T1: Day 2 | 3.2 (1.84)
  T1: Day 3 | 2.2 (1.61)
  T1: Day 4 | 2.5 (2.14)
  T1: Day 5 | 2.3 (2.21)
  T1: Day 8 | 2.5 (2.37)
  T1: Day 15 | 3.2 (2.48)
  T1: Day 28 | 3.4 (1.80)
  T2: Baseline (pre-dose): number analyzed (Participants) | 15
  T2: Baseline (pre-dose) | 5.4 (1.18)
  T2: Day 1: number analyzed (Participants) | 15
  T2: Day 1 | 5.2 (1.32)
  T2: Day 2: number analyzed (Participants) | 15
  T2: Day 2 | 3.5 (2.36)
  T2: Day 3: number analyzed (Participants) | 15
  T2: Day 3 | 1.9 (1.28)
  T2: Day 4: number analyzed (Participants) | 15
  T2: Day 4 | 2.1 (1.58)
  T2: Day 5: number analyzed (Participants) | 15
  T2: Day 5 | 1.9 (1.53)
  T2: Day 8: number analyzed (Participants) | 15
  T2: Day 8 | 2.2 (2.21)
  T2: Day 15: number analyzed (Participants) | 14
  T2: Day 15 | 2.4 (2.21)
  T2: Day 28: number analyzed (Participants) | 15
  T2: Day 28 | 2.9 (2.46)

5. Secondary Outcome: Change in Numeric Pain Rating Scale (NPRS) Scores for Back Pain From Baseline
Description: The NPRS is an 11-point scale (0- to 10-point scale where 0 is no pain and 10 is worst pain imaginable) that allows subjects to rate the severity of their pain intensity at various points in time (Turk et al., 2003). Subjects used the NPRS to record their current pain, average pain over 24 hours, and worst pain over 24 hours for both affected leg(s) and back pain. NPRS average back pain scores over 24 hours are presented.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SP-102
Number analyzed (Participants) | 19
score on a scale
  T1: Baseline (pre-dose) | 5.2 (1.46)
  T1: Day 1 | 5.2 (1.50)
  T1: Day 2 | 3.5 (2.14)
  T1: Day 3 | 2.3 (1.45)
  T1: Day 4 | 2.7 (2.11)
  T1: Day 5 | 2.6 (2.39)
  T1: Day 8 | 2.8 (2.48)
  T1: Day 15 | 3.2 (2.46)
  T1: Day 28 | 3.9 (1.90)
  T2: Baseline (pre-dose): number analyzed (Participants) | 15
  T2: Baseline (pre-dose) | 5.4 (1.35)
  T2: Day 1: number analyzed (Participants) | 15
  T2: Day 1 | 5.3 (1.35)
  T2: Day 2: number analyzed (Participants) | 15
  T2: Day 2 | 3.5 (2.33)
  T2: Day 3: number analyzed (Participants) | 15
  T2: Day 3 | 2.1 (1.55)
  T2: Day 4: number analyzed (Participants) | 15
  T2: Day 4 | 2.8 (1.81)
  T2: Day 5: number analyzed (Participants) | 15
  T2: Day 5 | 2.3 (1.35)
  T2: Day 8: number analyzed (Participants) | 15
  T2: Day 8 | 2.4 (2.03)
  T2: Day 15: number analyzed (Participants) | 14
  T2: Day 15 | 2.9 (1.96)
  T2: Day 28: number analyzed (Participants) | 15
  T2: Day 28 | 3.2 (2.27)

6. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events (TEAEs)
Description: Incidence of treatment-emergent AEs (TEAEs) related to study drug.
Time Frame: 12 weeks
Population: 19 subjects were enrolled and received an index (T1) injection of SP-102. 15 subjects received a (T2) injection of SP-102.
Measure: Number; unit: events
Arm/Group | SP-102
Number analyzed (Participants) | 19
events
  Treatment 1 | 20
  Treatment 2: number analyzed (Participants) | 15
  Treatment 2 | 10

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | SP-102
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 13/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SP-102 (N=19)
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Food poisoning (Gastrointestinal disorders) | 1
Gastrooesophageal refluxdisease (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 2
Blood glucose increased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 7
Migraine (Nervous system disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has the right to first publication of the results of the study. Following the first publication, PIs may publish study data or results; however, the proposed publication must be submitted to the Sponsor for review and approval in writing at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study Data.

DOCUMENTS (2):
  • Study Protocol (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT03613662/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT03613662/SAP_001.pdf